CLINICAL TRIAL: NCT05463692
Title: CAMELLIA Cohort: A Longitudinal Study to Understand Sexual Health and Prevention Among Women in Alabama
Acronym: CAMELLIA
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Lynn T. Matthews, Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 4662864; Accession Number:4662864 (Other: Health and Human Development)
Record Dates: First submitted 2022-07-13; First posted 2022-07-19 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Hiv; Sexually Transmitted Diseases
Keywords: HIV prevention education; STI prevention education; Pre-exposure prophylaxis (PrEP)
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm - CAMELLIA Cohort (Experimental): To better understand contextual factors among people who identify as women in Alabama that predict STI/HIV infection and PrEP use, we will refine an existing evidence-based mobile health app (HealthMpowerment or HMP) to optimally engage and retain a digital cohort of women at-risk for HIV infection (i.e. prior infection in the past 3 months with gonorrhea or syphilis). Using a sampling strategy based on geospatial analysis of HIV-risk, we will enroll and follow our factors associated with incident STI/HIV infection as well as utilization of PrEP through self-collected STI/HIV testing and survey assessments.
  Interventions: Behavioral: Camelia Cohort

INTERVENTIONS:
Behavioral: Camelia Cohort — Through the HealthMpowerment (HMP) app tailored for women, we will be able to provide informational content, access to resources, PrEP locators and additional gamification features to optimally engage and retain our cohort, which may support linkage to PrEP care.

SUMMARY:
Pre-exposure prophylaxis (PrEP) is an important biomedical human immunodeficiency virus (HIV) prevention tool and may particularly benefit black, cis and trans-gender women, who are at an increased risk for HIV and Sexually Transmitted Infections (STIs). The purpose of this study is to use a population-based approach to create a cohort of cis and trans-gender women at risk for future HIV acquisition to better understand the factors associated with the risk of STIs and HIV diagnosis and predictors of PrEP use.

DETAILED DESCRIPTION:
To better understand contextual factors among people who identify as women in Alabama that predict STI/HIV infection and PrEP use, we will refine an existing evidence-based mobile health app (HealthMpowerment or HMP) to optimally engage and retain a digital cohort of women at-risk for HIV infection (i.e. prior infection in the past 3 months with gonorrhea or syphilis). Using a sampling strategy based on geospatial analysis of HIV-risk, we will enroll and follow our cohort longitudinally to assess factors associated with incident STI/HIV infection as well as utilization of PrEP through iterative self-collected STI/HIV testing and survey assessments.

ELIGIBILITY:
Inclusion Criteria:

* Self identify as a Cis-gender or Trans-gender woman
* Age 18 - 89
* Reported STI in past 3 months by the Alabama Department of Public Health (ADPH)
* Gonorrhea and Syphilis negative
* HIV negative at screening encounter
* Live in Alabama
* Have access to a private smart phone

Exclusion Criteria:

* Live outside of Alabama
* Positive diagnosis for HIV, Gonorrhea, or Syphilis

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligible persons for screening include those who identify as women.
Enrollment: 830 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Annualized Sexually Transmitted Infections (STIs) | From time of enrollment through study completion at 24 months
  We will calculate incidence of gonorrhea and new positive cases of syphilis.

SECONDARY OUTCOMES:
Pre-Exposure Prophylaxis (PrEP) uptake | From time of enrollment through study completion at 24 months
  We will calculate incidence of PrEP initiation, as reported by participants and confirmed through medical record review or through Dried Blood Spot (DBS) sampling confirmed presence of tenofovir-base PrEP (TFV-dp).

CONTACTS AND LOCATIONS:
Overall Officials: Lynn T. Matthews, MD, MPH, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States